CLINICAL TRIAL: NCT04725396
Title: A Randomized Prospective Multicenter Study Comparing Fibula Free-flap Mandibular Reconstruction With or Without Preoperative Virtual Planning in Patients With Oral or Oropharyngeal Cancer
Brief Title: Study Comparing Fibula Free-flap MR With or Without PVP in Patients With OOPC
Acronym: CURVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UC-HNG-2009; 2020-A02655-34 (Registry Identifier: ANSM)
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Oropharynx Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma
Keywords: fibula free-flap; mandibular reconstruction; preoperative virtual planning
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Mandibular Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing PVP-assisted MR (Experimental): PVP is based on CT-scan with millimetric thin slice acquisitions of the facial bone and fibulas. The surgeon defines the exact sites of the intended mandibular osteotomies. A single external subcontracted laboratory (Materialise®) produces the various cutting guides for mandibular resection, flap conformation and the preformed plates for flap osteosynthesis. Flap conformation is entirely performed at the donor site before section of the vascular pedicle (flap still vascularized).
  Interventions: Device: Mandibular Reconstruction (MR) with Preoperative Virtual Planning (PVP).
- Patients undergoing conventional (i.e. without PVP) MR (Active Comparator): Flap modeling and positioning requires one or multiple cuneiform osteotomies. The bone transplant is shaped to restore the contours of the mandibular defect using preoperative imaging studies and the resection specimen. Flap conformation begins at the donor site and is generally completed at the recipient site after fibular pedicle section and before microvascular anastomosis (during ischemia time). The different bone fragments are fixed together and to the native mandible using either titanium miniplates or reconstruction plate and monocortical screws. Regardless of the material used for fixing the fibular flap to the native mandible, the use of a reconstruction plate adapted to the native mandible (or other similar techniques) prior to tumor resection is recommended to guide flap shaping and positioning, and to insure an accurate MR.
  Interventions: Device: Conventional Mandibular Reconstruction (MR without PVP)

INTERVENTIONS:
Device: Mandibular Reconstruction (MR) with Preoperative Virtual Planning (PVP). — PVP-assisted mandibular reconstruction includes the production of the surgical cutting guides required for mandibular resection and fibula free-flap conformation and of the preformed plates for flap osteosynthesis (for all patients, PVP will be done by the same laboratory).
  Arms: Patients undergoing PVP-assisted MR
Device: Conventional Mandibular Reconstruction (MR without PVP) — Conventional Mandibular Reconstruction
  Arms: Patients undergoing conventional (i.e. without PVP) MR

SUMMARY:
This is a national multicenter, randomized, stratified, open label study, aiming to compare mandibular reconstruction (MR) with or without preoperative virtual planning (PVP), in patients with oral/oropharyngeal cancer (OOPC).

DETAILED DESCRIPTION:
PVP-assisted MR includes the production of the surgical cutting guides required for mandibular resection and fibula free-flap conformation and of the preformed plates for flap osteosynthesis (for all patients, PVP will be done by the same laboratory: Materialise laboratory).

PVP-assisted MR includes the production of :

* surgical cutting guides required for mandibular resection and fibula free-flap conformation
* preformed plates for flap osteosynthesis

Patients will be selected after the multidisciplinary decision of oncological surgery including segmental mandibulectomy and immediate MR. Patients will be randomized in 2 groups (ratio 1:1, stratified on center and tumor N status [0-1 vs 2-3]).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over
2. Primary or recurrent OOPC, histologically proven, requiring segmental mandibulectomy
3. Planned immediate fibula free flap MR to be performed at the same time as the tumor ablation by segmental mandibulectomy
4. MR requiring at least one osteotomy for contouring the flap (i.e. at least 2 bone fragments)
5. East Cooperative Oncology Group (ECOG) performance status 0 or 1
6. American Society of Anesthesiologists Physical Status (ASA) score 1, 2, or 3
7. Patients considered fit for surgery as decided by the multidisciplinary team
8. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures
9. Patients must be affiliated to a Social Security System (or equivalent)
10. Patients must have signed a written informed consent form prior to any trial specific procedures. If the patients are physically unable to give their written consent, a trusted person of their choice, not related to the investigator or the sponsor, can confirm in writing the patient's consent

Exclusion Criteria:

1. Non resectable tumors (T4b primary tumor, non resectable metastatic lymph nodes)
2. Comorbidities factors that would contraindicate surgery (such as severe peripheral artery disease)
3. MR requiring no osteotomy for contouring the flap (i.e. one bone fragment)
4. Patients with distant metastatic disease as determined by routine pre-operative staging radiological investigations e.g. CT thorax and upper abdomen or positron emission tomography (PET)-CT
5. Other uncontrolled malignancy
6. Serious, non-healing or dehiscing wound, active ulcer or ongoing bone fracture at the free-flap donor site
7. Patients unwilling or unable to comply with the medical follow-up required by the trial because of psychosocial, familial, social, or geographical reasons
8. Participation in another clinical study with an investigational medicinal product during the last 30 days prior to inclusion
9. Patients deprived of their liberty or under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
General Oral Health Assessment Index (GOHAI) | 1-year
  Oral health-related quality of life (QoL) measured 1 year after surgery using the GOHAI in the 2 groups of patients (MR with or without PVP).
  The GOHAI is an oral-disease-specific QoL measure made by the patient. The GOHAI comprises 12 items grouped into three dimensions: the functional dimension (eating, speaking, swallowing); the pain or discomfort dimension (drugs, gingival sensitivity, discomfort when chewing certain foods); and, the psychosocial dimension (concerns, relational discomfort, appearance). The response format for each item is based on a five-point Likert scale: always = 1; often = 2; sometimes = 3; seldom = 4; never = 5. A summary score (ranging from 0 to 60) is calculated for each patient with a higher score indicating better oral health. GOHAI scores close to 30 have been reported in head and neck cancer patients after oncologic surgery and pedicled or free flap reconstruction.

SECONDARY OUTCOMES:
Time between randomization and surgery | At the time of surgery, up to 45 days after randomization
  Mean and median time between randomization and surgery
Total operative time and flap ischemia time | Post surgery, up to 45 days after randomization
  Mean and median total operative time and mean and median flap ischemia time
Postoperative surgical complication rate (including free-flap failure rate) | Post surgery, up to 45 days after randomization
  Surgical complication rates defined as local complication requiring another intervention in the first postoperative month, including free-flap failure rates
Delayed surgical complication rate | Post surgery, up to 45 days after randomization
  Delayed surgical complication rates defined as local complication occurring after the first postoperative month: non-union (pseudo-arthrosis), osteosynthesis-associated infection…
Functional outcome: Performance Status Scales for Head and Neck (PSS-HN) | At baseline and at 1 year
  The PSS-HN is a 3-item scale designed to evaluate functional performance of H&N cancer patients, specifically Normalcy of Diet, Eating in Public, and Understandability of Speech. Each subscale is rated based on semi-structured interview with a score of 0 to 100, with higher scores indicating better performance. The subscale scores are reported separately, and the Normalcy of Diet subscale will be the primary score of interest for this trial.
  The PSS-HN can be rated by health professionals including speech & language therapists and research nurses. The person collecting this data will remain consistent, as far as is feasible, throughout the course of the study. Scores are determined following an unstructured interview.
Functional outcome: Mouth opening range/capacity | At baseline and at 1 year
  Functional outcomes assessed by mouth opening range/capacity at baseline and at 1 year.
  It will be performed by using a caliper square to measure in millimeters the inter-incisor gap, assessed by the investigator.
Functional outcome: MD Anderson Dysphagia Inventory (MDADI) | 1 year
  The MDADI is a self-administered questionnaire designed specifically for evaluating the impact of dysphagia on the QoL of patients with head and neck cancer. It surveys QoL issues relevant to swallowing via several subscales: Emotional, Functional, and Physical. A fourth measurement, the Global subscale, is a single question designed to establish quickly an overall assessment that pertains to swallowing. A score ranging from 0 to 100 is calculated for each subscale, with higher scores indicating higher levels of dysphagia.
Functional outcome: Speech Handicap Index (SHI) | 1 year
  The SHI is a well-validated and widely used self-questionnaire for assessing speech problems in OOPC patients. It comprises 3 items and provides insight into the nature and severity of patients' complaints. Response categories for all but 1 item range on a 5-point scale (''never,'' ''almost never,'' ''sometimes,'' ''almost always,'' and ''always''). The questionnaire also includes an overall speech quality item, with 4 response categories (''good,'' ''reasonable,'' ''poor,'' and ''severe''). A total SHI score is calculated by summing all items (score range, 0-120), with higher scores indicating higher levels of speech related problems.
Functional dental status | At baseline and at 1 year
  Functional dental status (>6; 4-6, <4 functional dental units; type of dental rehabilitation) of the patients
Aesthetic outcome | 1 year
  Subjective assessment of the aesthetic outcome in the head and neck area using a visual analog scale (VAS) by the patient and the surgeon (assessed separately).
  The AESTHETIC VAS is a validated, subjective measure for esthetical perception. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "very poor looking"(0) and "very nice looking" (10).
Morphological results: mandibular angle | At 1 year
  Morphological results measured by the differences between the preoperative and postoperative measurements on 3D-CT-scan. The mandibular angle (in degrees) measured the amplitude of the angle existing between the ramus and body of the mandible.
Morphological results: bi-gonial diameter | At 1 year
  Morphological results measured by the differences between the preoperative and postoperative measurements on 3D-CT-scan. The bi-gonial diameter (in millimeter), a measure of the contracture/reduction of the arch, is intended to measure the preservation of the native mandibular arch anatomy.
Morphological results: position of the gnathion | At 1 year
  Morphological results measured by the differences between the preoperative and postoperative measurements on 3D-CT-scan. The lateral deviation (in millimeter) of gnathion in relation to the midsagittal plane will determined the degree of mandibular asymmetry.
Pain in the head and neck area | At 1 year
  "no pain" (0) and "worst pain" (10).
Evolution of patient QoL: GOHAI score | At baseline, at 6 months, and at 1 year
  Evolution of patient QoL GOHAI score at 6 months (this score will be compared to the score measured at baseline and at 1 year).
  The GOHAI is an oral-disease-specific QoL measure made by the patient. The GOHAI comprises 12 items grouped into three dimensions: the functional dimension (eating, speaking, swallowing); the pain or discomfort dimension (drugs, gingival sensitivity, discomfort when chewing certain foods); and, the psychosocial dimension (concerns, relational discomfort, appearance). The response format for each item is based on a five-point Likert scale: always = 1; often = 2; sometimes = 3; seldom = 4; never = 5. A summary score (ranging from 0 to 60) is calculated for each patient with a higher score indicating better oral health. GOHAI scores close to 30 have been reported in head and neck cancer patients after oncologic surgery and pedicled or free flap reconstruction.
Evolution of patient QoL: Quality of life questionnaire - Core 30 (QLQ-C30) score | At baseline, at 6 months and at 1 year.
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The EORTC QLQ-C30 is a general self-report questionnaire designed to assess QoL in cancer patients. It consists of five functioning scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea, and vomiting), a global QoL scale, and six single questions assessing additional symptoms commonly reported by cancer patients.
  As recommended by the EORTC, the scales and single-item variables of the QLQ-C30 will be linearly transformed into a score from 0 to 100. A high score for a functioning scale and for the global QOL scale represents a better level of functioning, whereas a high score for a symptom scale or a single item scale denotes a high level of symptoms or problems.
Evolution of patient QoL: Quality of Life Questionnaire - Head & Neck Cancer Module (QLQ-H&N35) score | At baseline, at 6 months and at 1 year.
  The EORTC QLQ-H&N35 is a tumor specific self-report questionnaire for head and neck cancer patients including seven symptoms scales (pain, swallowing, senses, speech, social eating, social contacts, and sexuality) and six single items (teeth problems, mouth opening, dry mouth, sticky saliva, coughing, and feeling ill).
  As recommended by the EORTC, the scales and single-item variables of the H&N35 questionnaire will be linearly transformed into a score from 0 to 100. A high score for a functioning scale and for the global QOL scale represents a better level of functioning, whereas a high score for a symptom scale or a single item scale denotes a high level of symptoms or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre BOZEC, Principal Investigator — Centre Antoine Lacassagne, Nice
Locations (10):
- France (10):
  - CHU Groupe Hospitalier Pellegrin, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - CHU Gui de Chauliac, Montpellier
  - CHU Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Pontchaillou, Rennes
  - IUCT-O, Toulouse
  - CHR de Valenciennes, Valenciennes
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No